CLINICAL TRIAL: NCT06484127
Title: Heterogeneity of Tertiary Lymphoid Structures Predicts Distinct Malignancy and Immune Microenvironment in Prostate Cancer: a Retrospective Cohort Study
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Wang Zhongyuan, Study Director, Fudan University
Other Study IDs: 050432-4-2307E
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- tertiary lymphoid structure positive patients
- tertiary lymphoid structure negative patients

SUMMARY:
The aim of this study was to reveal the predictive value of spatial heterogeneity and maturity difference of tertiary lymphoid structure in pathological sections of prostate cancer patients for clinical features and prognosis. It provides a new idea for the selection of prostate cancer immunotherapy population in the future.

ELIGIBILITY:
Inclusion Criteria:

1.patients diagnosed with prostate cancer who underwent radical prostatectomy or prostate puncture

Exclusion Criteria:

1. incomplete medical records, inadequate follow-up information, and confirmed non-prostatic acinar adenocarcinoma.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients diagnosed with prostate cancer who underwent radical prostatectomy or prostate puncture
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Correlation between the detection of TLS(tertiary lymphoid structure) and clinical features | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China